CLINICAL TRIAL: NCT03402815
Title: Efficacy of Maraviroc in Modulating Atherosclerosis in HIV Patients.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Of Perugia (Other)
Responsible Party: Principal Investigator, Elisabetta Schiaroli, Researcher, University Of Perugia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: UPerugia03
Record Dates: First submitted 2018-01-10; First posted 2018-01-18 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: HIV Infection With Other Conditions; Cardiovascular Risk Factor; Atherosclerosis; Inflammation
Keywords: HIV; Maraviroc; Atherosclerosis
MeSH Terms: conditions — Atherosclerosis; Inflammation | interventions — Maraviroc

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A (Experimental): Patients received Maraviroc 300 mg/day in addition to current ART for 24 weeks. At the end of the first 24-week period patients were switched to ART with no additional treatment.
  Interventions: Drug: Maraviroc 300 mg
- B (Experimental): Patients received ART with no additional treatment for 24 weeks. At the end of the first 24-week period patients were switched to Maraviroc 300 mg/day in addition to current ART.
  Interventions: Drug: Maraviroc 300 mg

INTERVENTIONS:
Drug: Maraviroc 300 mg — Patients were randomly allocated with an AB/BA cross over design to either maraviroc 300 mg/day to current ART for 24 weeks (A) or no additional treatment (B). At the end of the first 24-week period patients were switched to the alternative arm.

SUMMARY:
The investigator tested the efficacy of maraviroc intensification on down-regulating atherosclerotic progression in HIV infected patients with optimal viro-immunologic control and at high cardiovascular risk.

DETAILED DESCRIPTION:
Experimental CCR5 antagonism with maraviroc in atherosclerosis-prone mice and preliminary data in humans suggest an anti-atherosclerotic effect of the drug. The investigators assessed the impact of maraviroc treatment in HIV-infected patients on several subclinical indicators of atherosclerosis and putative mechanisms for such an effect.

HIV-treated patients under effective antiretroviral (ART) therapy, with a Framingham risk score >20% and a brachial flow-mediated dilation (bFMD) <4%, as indices of high cardiovascular risk, were recruited. Maraviroc (300 mg per os for 24 weeks) was administered on top of ART to all participants using a cross-over design. Brachial FMD, carotid-femoral pulse wave velocity (cfPWV) and carotid intima-media thickness (cIMT) were measured as non-invasive markers of atherosclerosis. Vascular competence, as expressed by the ratio of circulating endothelial micro-particles (EMPs) to endothelial progenitor cells (EPCs), as well as markers of systemic inflammation, monocyte activation and platelet activation were assessed.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients were consecutive ≥50-year-old individuals, treated for over 1 year with an effective protease inhibitor ART regimen (HIV RNA <50 copies/mL), with CD4 T cell counts > 300/ mm3 for at least 6 months and a Framingham risk score >20% and bFMD <4%.

Exclusion Criteria:

* Patients over 70 years of age, with life expectancy < 12 months, with known platelets functional defects or alcohol chronic abuse were excluded.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Change Flow Mediated Dilation | 24 weeks
Change in Intima-Media Thickness | 24 weeks
Change in carotid-femoral Pulse Wave Velocity | 24 weeks

SECONDARY OUTCOMES:
change in inflammatory markers | 24 weeks
  change in CRP, IL6, D-dimer
Endothelial microparticles/endothelial progenitor cells ratio | 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Elisabetta Schiaroli, Perugia, Italy